CLINICAL TRIAL: NCT05540366
Title: Effects of Aerobic Exercise on Pain in Patients With Myogenous Temporomandibular Disorders and Suspicion of Central Sensitization: A Pilot Randomized Controlled Trial
Brief Title: Effects of Aerobic Exercise on Pain in Patients With Myogenous Temporomandibular Disorders and Suspicion of Central Sensitization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Flora Dantony, Physical therapy department, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Flora Dantony
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Temporomandibular Disorder; Central Sensitisation; Myofascial Pain Syndrome; Endurance Training
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Exercise; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Myogenous temporomandibular subjects
  Physical therapy combined with aerobic exercise: 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions, combined with a 30 minutes aerobic exercise programme on a bike.
  Interventions: Other: Physical therapy combined with aerobic exercise
- Control group (Active Comparator): Myogenous temporomandibular subjects
  Physical Therapy: 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions (same programme than the intervention group)
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical therapy combined with aerobic exercise — 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions, combined with a 30 minutes aerobic exercise programme on a bike.
  Arms: Intervention Group
Other: Physical Therapy — 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions (same programme than the intervention group)
  Arms: Control group

SUMMARY:
Temporomandibular disorders are common in the general population, the myogenic subtype being the most frequent. Central sensitization seems to be present in this pathology, with a decreased pain pressure threshold observed in both local and remote areas. The best evidence-based treatment consists in combining education, manual therapy and therapeutic exercise in both temporomandibular and cervical regions. Aerobic exercise showed to be effective in subjects with chronic pain and central sensitization, by inducing an hypoalgesic effect. However, there isn't investigation about the effects of aerobic exercise in subjects with myogenic temporomandibular disorders and central sensitization. Thus, the aim of the pilot study is to determine if adding aerobic exercise to an effective physical therapy programme is more effective than physical therapy alone to improve pain pressure threshold in subjects with myogenic temporomandibular disorders and suspicion of central sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a myogenic temporomandibular disorder (DC/TMD) by an odontologist.
* A minimum score of 30 in the Central Sensitization Index
* Positive FRT

Exclusion Criteria:

* History of trauma, TMJ or cervical fracture the past three months
* History of TMJ or cervical surgery
* Systemic, rheumatic, metabolic, neurologic, psychiatric, pulmonary diseases or neoplastic malignant
* History of cardiovascular diseases which contraindicate aerobic exercise
* Current orthodontic treatment, splints for bruxism
* Drug addiction, alcoholism
* Pregnancy
* Use of analgesic medication less than 48 hours before each data collection
* Physical therapy treatment during the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of baseline in Pain Pressure Threshold at 2 weeks, 1 month (final) and 3 months (post) | Baseline - 2 weeks - 1 month (final) - 3 months
  Bilateral measure with digital algometer: TMJ, masseter, temporal, SCOM, achilles Tendon

SECONDARY OUTCOMES:
Change of baseline in Central Sensitization at 2 weeks, 1 month (final) and 3 months (post) | Baseline - 2 weeks - 1 month (final) - 3 months post
  Central Sensitization Index: 25 items, from 0 to 100 (0-29=subclinic; 30-39=mild; 40-59=moderate; 60-100=extrem)
Change of baseline in Pain intensity at 2 weeks, 1 month (final) and 3 months (post) | Baseline - 2 weeks - 1 month (final) - 3 months posts
  Visual Analog Scale: 100mm (no pain to worst pain)
Change of baseline in Jaw function at 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months post
  Fonseca Anamnestic Index. 10 questions with a three-point scale: 0 = no, 5 = sometimes and 10 = yes; total score from 0 good function, to 100 worst.
Change of baseline in Jaw range of motion al 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months posts
  Millimeter metalic rule to assess opening, lateral and protrusion jaw range of motion
Change of baseline in Cervical global ROM at 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months post
  CROM for global cervical range (flexion, extension, rotations, inclinations)
Change of baseline in Upper cervical ROM at 2 weeks, 1 month (final) and 3 months (post) | Baseline - 2 weeks - 1 month (final) - 3 months posts
  Assessment of upper cervical ROM performing the Flexion Rotation Test with a CROM device
Change of baseline in Neck disability at 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months posts
  Neck Disability Index: from 0 to 50 (0-4= no disability; 5-14=mild; 15-24=moderate; 25-34=severe; 35-50=complete)
Change of baseline in Anxiety and depression at 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months posts
  Hospital Anxiety and Depression Scale: 2 subscales, one for anxiety and the other one for depression. Each scale score is from 0 (less) to 21 (worst)
Change of baseline in Sleep Quality at 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months posts
  Pittsburgh Sleep Quality Index: maximum score of 21; 5 being the cut-off point.
Change of baseline in Perceived change at 1 month (final) and 3 months (post) | Baseline - 1 month (final) - 3 months posts
  Global Rating of Change scale: 15 points, from -7 (worst) to 7 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Spain

IPD SHARING:
Plan to Share IPD: No